CLINICAL TRIAL: NCT05734339
Title: Patient-Reported Outcomes of Benralizumab in Real-World Use in Severe Eosinophilic Asthma Patients in Taiwan
Brief Title: Patient-Reported Outcomes of Benralizumab in Real-World Use in Severe Eosinophilic Asthma Patients in Taiwan (BEAT)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00109
Record Dates: First submitted 2022-12-15; First posted 2023-02-17 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
An open-label, single-arm, non-interventional, prospective, multicenter study involving primary data collection within real-world settings for patients who receive benralizumab for treatment of severe uncontrolled eosinophilic asthma

DETAILED DESCRIPTION:
Benralizumab (Fasenra®) is a respiratory biologic agent targeting interleukin-5 (IL-5), an important member of the inflammatory cascade responsible for the pathogenesis of severe asthma. In 2019, Taiwan Food and Drug Administration (TFDA) approved benralizumab for the treatment of severe eosinophilic asthma (SEA). Since March 2020, benralizumab has been reimbursed by Taiwan National Health Insurance (NHI).

This prospective study (BEAT) aims to understand the use, effectiveness, and patient reported outcomes (PRO) of reimbursed benralizumab treatment in a real-world setting in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrolment in the study and treated with benralizumab according to Taiwan label and reimbursement criteria must meet ALL the following criteria:

1. Male or female patients ≥ 18 years of age (or ≥ 20 years of age for patients enrolled before January 1st, 2023, according to age of majority as defined by Taiwan regulations), with physician's confirmed diagnosis of severe uncontrolled asthma
2. Asthma requiring medium- or high-dose inhaled corticosteroid plus long-acting β-adrenoceptor agonist as maintenance treatment
3. Patients who have been prescribed but not yet initiated* treatment with reimbursed benralizumab (Fasenra®) according to the SmPC, prior to signed informed consent, and for whom the decision to prescribe this therapy is clearly separated from the physician's decision to include the patient in the current study. *Note: Treatment may be initiated (administration of first injection) at or after enrolment.

   Benralizumab Taiwan reimbursement criteria:
   * ≥ 2 acute exacerbations in the last 12 months, including at least 1 associated with emergency department (ED) visit or hospitalization; AND
   * At least 6 months of maintenance OCS use at ≥ 5 mg/day of prednisolone or equivalent dose; AND
   * Peripheral blood eosinophil ≥ 300 cells/μL in the last 12 months within the year before the initiation of benralizumab.
4. Provision of signed written informed consent form (ICF) indicating that they understand the purpose of the study and procedures required for participation
5. Patients must be able and willing to read, comprehend written instructions, and complete the paper questionnaires required by the protocol (ACQ-5, PGI-C, and PGI-S).

In case a patient does not own a smartphone or is not willing to perform the home spirometer, enrolment into the study is up to the physicians' discretion. We anticipate that 90% of patients will participate the home spirometer assessment.

Exclusion Criteria:

Subject must not meet ANY exclusion criteria:

1. Documented active lung diseases other than asthma and not within reimbursed label
2. Currently enrolled in an interventional clinical study in parallel, except:

   * Patients being in parallel documented in a national asthma registry
   * Patients having completed any other clinical trials including those with biologic treatment.
3. An acute or chronic condition that, in the investigator's opinion, would limit the patients' ability to complete questionnaires, participate in this study, or impact the interpretations of results.
4. Concurrent biologics for asthma are not allowed. Acceptable wash-out periods for other asthma biologics: ≥ 30 days from last dose of previous biologics.
5. Patients already started benralizumab treatment are not allowed. If the patients had received benralizumab treatment before, there should be an interval of ≥ 6 months from the last dose of prior benralizumab course to the newly initiated benralizumab treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will recruit 57 adult patients with confirmed SEA who meet all inclusion criteria and none of the exclusion criteria. Approximately 8 hospitals will participate in the study which have experience with biologic treatment, can initiate treatment with benralizumab, and have a good oversight on the severe asthma population.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the change in asthma control after initiation of benralizumab in a real-world Taiwan setting | after 8 weeks of benralizumab treatment
  Primary outcome measure:
  Changes from baseline in Asthma Control Questionnaire, five-question version (ACQ-5)
  scored from 0 (totally controlled) to 6 (severely uncontrolled)
To evaluate the change in asthma control after initiation of benralizumab in a real-world Taiwan setting | after 1, 2, 3, 4, 24, and 56 weeks of benralizumab treatment
  Secondary outcome measure:
  Changes from baseline in ACQ-5
  scored from 0 (totally controlled) to 6 (severely uncontrolled)
To evaluate the change in asthma control after initiation of benralizumab in a real-world Taiwan setting | at 1, 2, 3, 4, 8, 24, and 56 weeks compared to baseline
  Secondary outcome measure:
  Percentage of patients with an improvement of ≥ 0.5 points (minimal clinically importance differences [MCID]) in ACQ-5
  scored from 0 (totally controlled) to 6 (severely uncontrolled)
To evaluate the change in asthma control after initiation of benralizumab in a real-world Taiwan setting | at 1, 2, 3, 4, 8, 24, and 56 weeks of benralizumab treatment
  Percentage of patients with well-controlled asthma (ACQ-5 ≤ 0.75), partly controlled asthma (ACQ-5 between > 0.75 and < 1.5) and not well-controlled asthma (ACQ-5 ≥ 1.5)
  scored from 0 (totally controlled) to 6 (severely uncontrolled)

SECONDARY OUTCOMES:
To assess change in overall asthma status and disease severity after initiation of benralizumab | at Week 1, 2, 3, 4, 8, 24, and 56 in asthma
  Patient Global Impression of Change (PGI-C) response and PGI-C responder endpoint (a little better, moderately better, much better)
  The PGI-C is a single item designed to capture the participant's perception in change in overall disease status since the first dose of benralizumab using a 7-point scale (1- much better to 7- much worse)
To assess change in overall asthma status and disease severity after initiation of benralizumab | Changes from baseline after 1, 2, 3, 4, 8, 24, and 56 weeks
  Patient Global Impression of Severity (PGI-S) in asthma
  The PGI-S is a single question designed to capture patient's perception of overall symptom severity on a scale of no symptom to very severe
To determine the change on lung function after treatment with benralizumab | after 24 and 56 weeks of treatment with benralizumab
  Pre-bronchodilator changes in FEV1 and FVC assessed by standard hospital spirometry (if available)
To assess the rate and change of acute exacerbations after initiation of benralizumab in a real-world Taiwan setting | from baseline at Week 24 and 56
  Annualized acute exacerbation rate and changes
To assess the rate and change of acute exacerbations after initiation of benralizumab in a real-world Taiwan setting | at Week 24 and 56
  Proportion of patients with 0, 1, and ≥ 2 acute exacerbations
To assess the rate and change of acute exacerbations after initiation of benralizumab in a real-world Taiwan setting | at Week 24 and 56
  Severity of exacerbation (use or temporary increase of systemic corticosteroids, emergency department visit, or hospitalization)
To assess the ability to reduce OCS dose after initiation of benralizumab in a real-world Taiwan setting | at Week 4, 8, 24, and 56
  Mean and median OCS daily dose reductions
To assess the ability to reduce OCS dose after initiation of benralizumab in a real-world Taiwan setting | at Week 4, 8, 24, and 56
  Proportion of patients with a ≥ 25%, ≥ 50%, ≥ 75%, and 100% OCS daily dose reduction
To assess the ability to reduce OCS dose after initiation of benralizumab in a real-world Taiwan setting | at Week 4, 8, 24, and 56
  Changes from baseline in cumulated OCS dose
To describe characteristics of patients with benralizumab treatment in a real-world Taiwan setting | known at the time of baseline data collection
  Baseline asthma disease history and commodities
To describe characteristics of patients with benralizumab treatment in a real-world Taiwan setting | at baseline and at Week 4, 8, 24, and 56
  Background medication
To describe characteristics of patients with benralizumab treatment in a real-world Taiwan setting | at baseline and Week 4, 8, 24, and 56
  Biomarker status (blood eosinophil and serum IgE level, if available)
To describe characteristics of patients with benralizumab treatment in a real-world Taiwan setting | through study completion, up to 56 weeks
  Adherence to benralizumab scheduled dose during study period and investigator-chosen reasons for discontinuation
To describe characteristics of patients with benralizumab treatment in a real-world Taiwan setting | in the past 12 months
  Most recent pre-bronchodilator FEV1 and FVC assessed by standard hospital spirometry

OTHER OUTCOMES:
To determine the clinical utility of home spirometer in severe asthma patient management in a real-world Taiwan setting | at Week 8, Week 24 and 56
  Correlation of ACQ-5 and FEV1 changeand long term-outcome (ACQ-5, FEV1, annualized exacerbation rate, OCS reduction)
To determine the clinical utility of home spirometer in severe asthma patient management in a real-world Taiwan setting | at baseline, Week 24 and 56
  Correlation between home spirometer and standard spirometry
To determine the clinical utility of home spirometer in severe asthma patient management in a real-world Taiwan setting | weekly from Week 1 to 4 and monthly from Week 8 to 56 during the treatment with benralizumab
  Pre-bronchodilator changes in FEV1 assessed by home spirometer ("MIR" Spirobank Smart)
To determine the clinical utility of home spirometer in severe asthma patient management in a real-world Taiwan setting | weekly from Week 1 to 4 and monthly from Week 8 to 56 during the treatment with benralizumab
  Pre-bronchodilator changes in FVC assessed by home spirometer ("MIR" Spirobank Smart)
To determine the clinical utility of home spirometer in severe asthma patient management in a real-world Taiwan setting | weekly from Week 1 to 4 and monthly from Week 8 to 56 during the treatment with benralizumab
  Pre-bronchodilator changes in PEF assessed by home spirometer ("MIR" Spirobank Smart)

CONTACTS AND LOCATIONS:
Overall Officials: Clara Tsai, Study Director — AstraZeneca
Locations (6):
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home